CLINICAL TRIAL: NCT04675450
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of n-Butylphthalide (NBP) Softgel Capsules Administered to Patients With Metastatic Breast Cancer to Prevent Nab-paclitaxel Induced Toxic Neuropathy
Brief Title: NBP in Women With Metastatic Breast Cancer to Prevent Nab-paclitaxel Induced Toxic Neuropathy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Further preclinical development activities required to proceed
Sponsor: Conjupro Biotherapeutics, Inc. (Industry)
Collaborators: CSPC-NBP Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CPO-NBP-2002
Record Dates: First submitted 2020-11-20; First posted 2020-12-19 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer; Peripheral Neuropathy
MeSH Terms: conditions — Breast Neoplasms; Peripheral Nervous System Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Interventions: Placebo (NBP placebo softgel capsules, 0 mg NBP, BID)
  Interventions: Drug: Placebo
- NBP (Active Comparator): Interventions: 800 mg NBP softgel capsules daily (400 mg BID)
  Interventions: Drug: NBP Softgel Capsules

INTERVENTIONS:
Drug: Placebo — Take 4 capsules BID on an empty stomach at least 1 hour before food intake, and remain fasting at least 1 hour after dosing
  Other Names: NBP Placebo Softgel Capsules
  Arms: Placebo
Drug: NBP Softgel Capsules — Take 4 capsules BID on an empty stomach at least 1 hour before food intake, and remain fasting at least 1 hour after dosing.
  Other Names: NBP
  Arms: NBP

SUMMARY:
Phase 2, randomized, double-blind, Placebo-Controlled, Multiple Dose Study for the treatment of Patients with Metastatic Breast Cancer.

DETAILED DESCRIPTION:
This is a multiple center, randomized, double-blind, Phase 2 study of NBP administered to women with metastatic breast cancer who receive nab-paclitaxel as therapy. Nab-paclitaxel will be administered at a dose >260 mg/m2 every 3 weeks for 4 planned cycles. Subjects will begin receiving NBP orally at a dose of 400 mg administered every 12-hours (BID) or matching placebo 5 days (10 doses) prior to starting nab-paclitaxel therapy and continue to self-administer it BID until Visit 6/Day 100/Week 15. The primary objective is to evaluate the efficacy of NBP relative to placebo at preventing or reducing symptoms associated with nab-paclitaxel induced toxic neuropathy (CIPN). The secondary objectives include an evaluation the efficacy of NBP relative to placebo at preventing or attenuating taxane induced acute pain syndrome (TAPS), the evaluation of the safety and tolerability of NBP relative to placebo and to determine if NBP administration impacts the pharmacokinetics of nab-paclitaxel or if nab-paclitaxel affects the pharmacokinetics of NBP.

ELIGIBILITY:
Inclusion Criteria

Subjects are eligible to participate in the study only if all the following criteria apply:

1. Women aged ≥18 and ≤75 years.
2. Pathologically confirmed metastatic breast cancer.
3. Are candidates for initial therapy with nab-paclitaxel, at a dose of >260 mg/m2 every 3 weeks for 4 planned cycles.
4. Concomitant antitumor drugs used to treat the underlying malignancy, including immunotherapies, other than nab-paclitaxel will be allowed.
5. Eastern Cooperative Oncology Group (ECOG) performance status scores of 0 - 2.
6. Life expectancy ≥6 months.
7. Women of childbearing potential (WOCBP) must have a negative serum human chorionic gonadotropin (HCG) pregnancy test at Screening and be practicing a medically acceptable method of contraception with an annual failure rate of less than 1% until the completion of the trial or 30 days after discontinuation of study treatment. Women are considered not childbearing if they are >1 year postmenopausal or surgically sterile (ie, hysterectomy, bilateral oophorectomy, or bilateral salpingectomy tubal ligation).
8. Able to complete study questionnaires by themselves or with assistance.
9. Capable of understanding the purpose and risks of the study and able to provide informed consent by signing the informed consent form.
10. Able to swallow softgel capsules as determined by the investigator.
11. Able to comply with all study requirements. Exclusion Criteria

Subjects are excluded from the study if any of the following criteria apply:

1. Non-metastatic breast cancer.
2. Subjects who are pregnant, lactating/breast-feeding, or plan to become pregnant within the next 3 months.
3. History of poorly controlled diabetes mellitus (hemoglobin A1C >8.0 at the time of the Screening visit).
4. History of fibromyalgia.
5. History of any signs or symptoms suggestive of neuropathy within 30 days of Screening as determined by the investigator based on the neurological examination.
6. History of taking any neurotoxic drugs within 6 months of Screening.
7. Current use of drugs that are used to treat neuropathic pain (eg, gabapentin, pregabalin, and duloxetine) within 30 days of Screening.
8. Current diagnosis of malignancy other than breast cancer.
9. Absolute neutrophil count <1.5 x 109 cells/L.
10. Platelet count <100,000 x 109/L.
11. Hemoglobin level <9 g/dL at Screening without transfusion (transfusion independent).
12. Corrected QTcF >470 msec (single tracing) at Screening and prior to randomization.
13. Chronic renal or hepatic disease.
14. Clinically significant renal dysfunction including serum creatinine level >1.5 mg/dL or calculated creatinine clearance ≥50 mL/minute at Screening.
15. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level >2.0 x upper limits of normal (ULN), or a bilirubin >1.5 x ULN unless in the setting of known Gilbert's disease at Screening.
16. History of HIV, hepatitis B, hepatitis C, or tuberculosis.
17. Major surgical procedures ≤30 days prior to starting study drug, or minor surgical procedures ≤7 days prior to starting study drug.
18. History of alcohol or drug dependence or is known to have abused alcohol within 30 days prior to screening.
19. Unwilling to abstain from alcohol and recreational drugs (with exception for medical marijuana) throughout the duration of participation in the study.
20. Positive urine drug screen at Screening (with exception for medical marijuana which is allowed).
21. Known hypersensitivity to celery or soybeans.
22. Known serious hypersensitivity to paclitaxel
23. Received treatment with any other investigational drug within 30 days before screening, was previously treated with NBP, is currently taking celery seed extract, or is currently participating in another clinical study
24. Any other reasons that in the opinion of the investigator make the subject unsuitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06-30 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Mean Change from Baseline in EORTC Quality of Life Questionnaire Chemotherapy-Induced Peripheral Neuropathy (EORTC QLQ-CIPN20) Sensory Subscale | Baseline and weeks 5, 8, 11 and 15
  Change from baseline in the mean EORTC QLQ-CIPN20 sensory subscale (converted to a 0-100 scale) collected during the treatment period at weeks 5, 8, 11 and 15.

SECONDARY OUTCOMES:
Number of Participants Requiring Rescue Medication | 15 weeks
  The number and percentage of participants requiring oxycodone of any amount anytime during the 15 week treatment period.
Days Free of Rescue Medication | 15 weeks
  The mean cumulative number of days free of oxycodone of any amount anytime for each participant during the 15 week treatment period.
Mean Change from Baseline in the Brief Pain Inventory Short Form (mBPI-SF) score. | 15 weeks
  The mean change from baseline (mean days 2-7 after first dose of NBP or Placebo) in the mBPI-SF total score to mean of all post-nab-paclitaxel mBPI-SF scores collected on days 2-7 after each of 4 nab-paclitaxel administration at days 7, 28, 49 and 70 during the 15 week treatment period.
Number of Participants with Treatment-Emergent Adverse Events | 19 weeks
  The number and percentage of participants with treatment-emergent adverse events according to MedDRA system organ class and preferred term with onset during the 15 week treatment period or 4 week follow-up.
Area Under the Curve (AUC) for NBP | 0, 1.5, 3, 4, 6, 8 and 24 hours - Days 6 and 7
  The AUC (h*ng/mL) be calculated using Phoenix WinNonlin software
Cmax for NBP | Time Frame: 0, 1.5, 3, 4, 6, 8 and 24 hours - Days 6 and 7
  Cmax (ng/mL) be calculated using Phoenix WinNonlin software
Tmax for NBP | 0, 1.5, 3, 4, 6, 8 and 24 hours - Days 6 and 7
  Tmax (hr) be calculated using Phoenix WinNonlin software
Area Under the Curve for Paclitaxel | 0, 1.5, 3, 4, 6, 8 and 24 hours - Days 6 and 7
  AUC (h*ng/mL) be calculated using Phoenix WinNonlin software
Cmax for Paclitaxel | 0, 1.5, 3, 4, 6, 8 and 24 hours - Days 6 and 7
  Cmax (ng/mL) be calculated using Phoenix WinNonlin software
Tmax for Paclitaxel | Time Frame: 0, 1.5, 3, 4, 6, 8 and 24 hours - Days 6 and 7
  Tmax (hr) be calculated using Phoenix WinNonlin software

CONTACTS AND LOCATIONS:
Overall Officials: Qingxi Wang, PhD, Study Director — Conjupro Biotherapeutics, Inc.